CLINICAL TRIAL: NCT01702701
Title: Eosinophilic Esophagitis Treatment: Montelukast vs Fluticasone
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCWEoEMVF
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2016-01

CONDITIONS: Eosinophilic Esophagitis; Dysphagia
MeSH Terms: conditions — Eosinophilic Esophagitis; Deglutition Disorders | interventions — montelukast; Fluticasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Active Comparator): patients will receive 10 mg po montelukast daily for 12 weeks.
  Interventions: Drug: Montelukast
- Fluticasone (Active Comparator): patients will receive 440mcg fluticasone po bid for 12 weeks
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Montelukast — montelukast 10mg po pill q day for 12 weeks
  Other Names: Singulair
  Arms: Montelukast
Drug: Fluticasone — fluticasone 440mcg po q bid x 12 weeks
  Other Names: Flovent
  Arms: Fluticasone

SUMMARY:
This study will compare response to treatment of Eosinophilic Esophagitis with montelukast vs standard therapy fluticasone. Investigators hypothesize that montelukast is equally effective in treating symptoms and histology of EoE when compared to fluticasone. The study will be conducted at multiple sites with Medical College of Wisconsin as the coordinating site. After identification and recruitment all patients will be randomized (provider blinded) to one of two medications: montelukast 10mg po qday vs fluticasone 440mcg po bid. Patients will also complete a pretreatment, 6 week therapy and 12 week therapy questionaire. They will then undergo a repeat endoscopy to evaluate endoscopic and histologic response.

DETAILED DESCRIPTION:
Eosinophilic esophagitis is an allergic condition of the esophagus with an incidence that is on the rise, and has limited treatment options. Current gold standard of treatment is with topical steroids (swallowed fluticasone). There is preliminary data that oral montelukast may prove to be effective in inducing and maintaining symptomatic along with histologic remission of this disease. Investigators will be comparing the effectiveness of singulair to swallowed fluticasone in inducing and maintaining histologic and symptomatic remission of eosinophilic esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of EoE on biopsy
* with >15 eos per HPF
* ages >18
* Both male and Female.
* Not pregnant

Exclusion Criteria:

* pregnancy
* patients receiving ongoing medical therapy for EoE
* patients who underwent dilation in the last 12 weeks with improvement in symptoms
* LA grade B or worse erosive esophagitis.
* age < 18
* nursing mothers
* use of prohibited concomitant medications : budesonide-oral compounded liquid, fluticasone or montelukast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Improvement in Dysphagia symptom score | 3 month

SECONDARY OUTCOMES:
Improvement in esophageal histology counts of eosinophils/hpf | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Walter Hogan, MD, Principal Investigator — Medical College of Wisconsin; Nikhil Shastri, MD, Study Director — Medical College of Wisconsin
Locations (2):
- United States (2):
  - GI Associates, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin